

# Protocol Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy and Safety of REL-1017 Monotherapy for Major Depressive Disorder (The RELIANCE-III Study)

Protocol Number: REL-1017-303

NCT Number NCT05081167

Name of Investigational Product: REL-1017

Phase of Development: 3

Indication: Major Depressive Disorder Sponsor: Relmada Therapeutics Inc.

Protocol Date: August 03 2022

Certain information within this protocol has been redacted to protect either personally identifiable information or company confidential information.

This may include, but is not limited to, redaction of the following:

- Names, addresses, and other personally identifiable information
- Proprietary information, such as scales or coding systems, which are considered confidential information.
- Other information as needed to protect the trade secret and/or confidential information of Relmada Therapeutics



# Protocol Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy and Safety of REL-1017 Monotherapy for Major Depressive Disorder (The RELIANCE-III Study)

Protocol Number: REL-1017-303

Name of Investigational Product: REL-1017

Phase of Development: 3

Indication: Major Depressive Disorder

Relmada Therapeutics, Inc.

Sponsor: 2222 Ponce de Leon Blvd, Floor 3

Coral Gables, FL 33134

Protocol Version:

Amendment Version:

Protocol Date: 03Aug2022

#### -CONFIDENTIAL-

This document and its contents are the property of and confidential to Relmada Therapeutics, Inc. Any unauthorized copying or use of this document is prohibited.

### PROTOCOL APPROVAL SIGNATURES

| Protocol Title: | A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled<br>Study to Assess the Efficacy and Safety of REL-1017 Monotherapy for<br>Major Depressive Disorder (The RELIANCE-III Study) |
|---|---|
| Protocol Number: | REL-1017-303 |
| <b>Protocol Version</b> | |
| Amendment Version | |
| AND AND ADDRESS OF THE PARTY OF | ucted in compliance with the clinical study protocol (and amendments), or Harmonisation (ICH) guidelines for current Good Clinical Practice egulatory requirements. |
| Sponsor Signatory | |
| Relmada Therapeutics | Signature |
| | Date (DD-Mmm-YYYY) |

#### INVESTIGATOR SIGNATURE PAGE

Protocol Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled

Study to Assess the Efficacy and Safety of REL-1017 Monotherapy for

Major Depressive Disorder (The RELIANCE-III Study)

**Protocol Number:** REL-1017-303

### Confidentiality and Current Good Clinical Practice (GCP)/E6(R2):

I agree, as an Investigator conducting this study:



| Name | Investigator Signature |
|-------------|------------------------|
| Title | Date (DD-Mmm-YYYY) |
| Institution | |

### 1 SYNOPSIS

| Title of Study | Study to Assess | icenter, Randomized, Double-Blind, Placebo-Controlled<br>the Efficacy and Safety of REL-1017 Monotherapy for<br>we Disorder (The RELIANCE-III Study) |
|---|---|---|
| Sponsor | Relmada Therapeutics, Inc. (Relmada) | |
| Investigators/Study Sites | Approximately | planned in the United States |
| Phase of Development | 3 | |

| Objectives | Endpoints |
|---|---|
| Primary | |
| | Absolute change from Baseline to Day 28 of the MADRS10 total score in REL-1017 compared to placebo Key Secondary Efficacy Endpoints |

# **Objectives Endpoints** Withdrawal Withdrawal Endpoints Signs and symptoms of withdrawal in approximately the first 200 completers of the 28-day double-blind treatment period during 14 days after last dosing: Withdrawal Objectives To evaluate signs and symptoms of withdrawal in approximately the first 200 participants, who complete the 28-

| Objectives | Endpoints |
|---|---|
| day double-blind treatment period, during 14 days after last dosing. | <ul> <li>Change from Day 28 until Day 42 in Clinical Opiate Withdrawal Scale (COWS) score</li> <li>Change from Day 28 until Day 42 in Subjective Opiate Withdrawal Scale (SOWS) score</li> <li>Change from Day 28 until Day 42 in Physician Withdrawal Checklist (PWC-20) score</li> </ul> |
| Safety | |
| To evaluate safety and tolerability of REL-1017 | <ul> <li>Treatment-emergent adverse events (TEAEs)</li> <li>Vital signs and weight</li> <li>Physical examination</li> <li>Clinical laboratory parameters (chemistry, hematology, and urinalysis)</li> <li>Columbia-Suicide Severity Rating Scale (C-SSRS)</li> <li>Global COVID-19 impact scale</li> </ul> |
| Pharmacokinetic Pharmacokinetic Objectives To evaluate pharmacokinetics (PK) of REL-1017 and potential metabolites | Pharmacokinetic Endpoints • Estimation of REL-1017 PK profile (maximum concentration [C <sub>max</sub> ], trough concentration [C <sub>trough</sub> ], and terminal half-life at steady state [t <sub>1/2</sub> ] based on sparse PK sampling |

| Stady Design | This is an outpatient, 2-arm, Phase 3, multicenter, randomized, double-<br>blind, placebo-controlled study to assess the efficacy and safety of<br>REL1017 at 25 mg once daily (QD) as monotherapy treatment for MDD |
|---|---|
| Investigational | REL-1017 in 25 mg and matching placebo |

| Due due d'Defeuer es Due de et | |
|---|---|
| Product/Reference Product | |
| Study Drug, Dose Schedule, and Mode of | REL-1017 in a 25 mg tablet for oral administration by mouth (PO) |
| Administration | The following dose schedule will be used in the study: |
| | Day 1 – loading dose: Three REL-1017 25 mg tablets (75 mg total) administered at the clinical study site, or Three matching placebo tablets administered at the clinical study site |
| | <ul> <li>Day 2 to Day 28 – maintenance dose:</li> <li>One REL-1017 25 mg tablet QD, or</li> <li>One matching placebo tablet QD</li> </ul> |
| Study Population and<br>Duration of Participation | Dosing should take place once daily at the same time each day. Adult participants (aged 18 to 65 years, inclusive) diagnosed with MDD (based on Structured Clinical Interview for DSM-5 [SCID-5] for MDD, matching Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition [DSM-5]), who are currently in a major depressive episode (MDE), The maximum duration of the MDE must not exceed 12 months. |
| | After signing of the informed consent form (ICF), each participant will |
| | undergo Screening Period of up to 30-days followed by a 28-day randomized double-blind placebo-controlled period, for a total of approximately 58 days of study participation. |

| | All participants who complete the 28-day treatment period will be offered the opportunity to enroll into a 1 year open-label study under its separate study protocol. Those participants who do not elect to enter the open-label study will return to the clinic up to 14 days after their final dose of study drug for final safety and study evaluations. |
|---|---|
| Planned Sample Size | The REL-1017-303 study is designed to achieve 90% power, with an overall two-tailed $\alpha$ -level of 0.05. |
| Inclusion Criteria | To enroll in the clinical study, participants must meet the following inclusion criteria: 1. Must be able to read, speak, and understand English or Spanish and must provide written informed consent prior to the initiation of any protocol-specific procedures. 2. Male or female participants, aged 18 to 65 years, inclusive. 3. Participant is willing and able to commit to meet all study requirements, adhere to the study drug regimen, and complete all assessments and all scheduled visits, per Investigator judgment. 5. Women of childbearing potential (WOCBP) and men whose sexual partners are WOCBP must use at least 1 highly effective method of contraception from Screening and for at least 2 months after the last study drug administration. Men and women must agree to abstain from sperm and egg donation, respectively, from Screening until at least 2 months after the last dose of study drug administration. For men with female sexual partners of childbearing potential, examples of medically acceptable forms of contraception include vasectomy or male condom for participants, plus an additional method of contraception for their female partners. Highly effective methods of contraception are those which have a failure rate of <1% (when implemented consistently and correctly) and include: |

- Intrauterine device (IUD)
- Bilateral tubal ligation, bilateral salpingectomy, or bilateral tubal occlusive procedure
- Hormonal contraceptives (i.e., oral, patch, or injectable)
- A double-barrier protection method (i.e., condom, sponge, or vaginal diaphragm with spermicide cream, foam, or gel)
- Abstinence from heterosexual intercourse is accepted if this is the participant's usual lifestyle and must be continued until at least 2 months after the last dose of study drug.

Women who are not of childbearing potential must be congenitally or surgically sterile (hysterectomy and/or bilateral oophorectomy/salpingo-oophorectomy, as determined by the participant's medical history) or must be post-menopausal. Post-menopausal is defined as being amenorrheic for at least 1 year without another cause and a follicle-stimulating hormone (FSH) level ≥40 mIU/mL as confirmation.

- Diagnosed with MDD as defined by the Diagnostic and Statistical Manual, Fifth Edition (DSM-5), and confirmed by the SCID-5 MDD.
- 7. Hamilton Depression Rating Scale-17 (HAMD17) score at Screening and independently confirmed by SAFER assessment.



#### **Exclusion Criteria**

- History or presence of clinically significant abnormality as assessed by physical examination, medical history, 12-lead ECG, vital signs, or laboratory values, which in the opinion of the Investigator would jeopardize the safety of the participant or the validity of the study results, including established QT prolongation, long QT syndrome, torsades de pointes, bradyarrhythmia, ventricular tachycardia, uncompensated heart failure (greater than New York Heart Association [NYHA] Class 1 congestive heart failure [CHF]), uncontrolled hypokalemia, or uncontrolled hypomagnesemia.
- More than class 2 angina pectoris or a myocardial infarction (MI) or acute coronary syndrome within the past 3 months.
- Any medical, psychiatric condition, or social context that, in the
  opinion of the investigator, is likely to unfavorably alter the riskbenefit of subject participation, to interfere with protocol compliance,
  or to confound safety or efficacy assessments.
- 4. Have any significant illness, of any nature, including possible Coronavirus-SARS-2 related fever and symptoms, requiring

- hospitalization, emergency treatment, or isolation (quarantine) within 4 weeks prior to Screening or during the Screening period, and as determined by the Investigator.
- 5. History or first degree relative with history of unexplained sudden death or long QT syndrome.
- 6. Triplicate 12-lead ECG with average QTcF (QT interval with Fridericia correction) ≥450 msec and/or a QRS interval ≥120 msec at Screening.
- 7. Current or recent uncontrolled orthostasis or orthostatic hypotension necessitating treatment.
- 8. Poorly controlled diabetes as defined by a glycosylated hemoglobin (HbA1c) >7.5%, despite standard care.
- Any use of long-term prescribed opioids (i.e., >120 days in a 6-month period) within 6 months prior to Screening or any recreational use of opioids.
- 12. Use of any antidepressant medication within 30 days prior to Screening and/or more than 1 antidepressant medication to treat the current MDE.
- 13. Use of any antipsychotic, anticonvulsant/antiepileptic, mood stabilizer, or stimulant medications within 30 days prior to Baseline.
- 14. Use of St. John's wort within 30 days prior to Baseline.
- 15. Participated in a ketamine, esketamine, dextromethorphan or any other NMDAR-antagonist study, or who received esketamine at any time.
- 16. Received ketamine, memantine, and/or dextromethorphan treatment within 30 days prior to Screening.
- 17. History of allergy or hypersensitivity to methadone or related drugs.
- 18. Receiving new-onset psychotherapy (individual, group, marriage, or family therapy) within 2 months prior to Screening, or planning to start psychotherapy at any time during participation in the study.
- 19. Any lifetime experience of electroconvulsive therapy (ECT) and/or vagus nerve stimulation (VNS), or any other type of physical brain stimulation.
- 20. Received repetitive transcranial magnetic stimulation (rTMS) less than 6-months prior to the Screening visit.
- 21. Any current psychiatric disorder (i.e., a condition that is the primary focus of distress and/or treatment other than MDD), as defined by the DSM-5 and confirmed by psychiatric history and/or examination by the Investigator. These disorders include, but are not limited to, any psychotic disorder, post-traumatic stress disorder, borderline personality disorder, antisocial personality disorder, obsessive-compulsive disorder, intellectual disability, or pervasive developmental disorder.
- 22. Participants who, in the Investigator's judgment, are at significant risk for suicide. A participant with a C-SSRS ideation score of 4 or 5 within the last 6 months or any suicide attempt within the past year of either Screening or Baseline must be excluded.
- 23. Any lifetime history of bipolar I or II disorder, psychosis and/or mania



# Study analysis populations will be defined as follows: Statistical Data Analysis Screened / Randomized / Enrolled Set: The Screened/Enrolled Set will include all participants who signed an informed consent. The Randomized Set will include all participants randomized, and will be used for the presentation of participants in all listings. Full Analysis Set (FAS): Participants who are randomized and dosed, irrespective of any deviation from the protocol or premature discontinuation. Participants will be analyzed according to randomized treatment. The FAS will be used as primary population for analyses of efficacy estimands and endpoints. Per-Protocol Set: Valid completer, i.e., participants who complete the 28day treatment and do not have any major protocol deviations impacting the efficacy assessments. This set will be analyzed according to the treatment actually received. Safety Set: All randomized participants who received any dose of study drug. The treatment group assignment in this population will be according to the treatment received. This population will be used for the analysis of safety. **Pharmacokinetic (PK) Set:** All participants who received at least one dose of REL-1017 and have at least one PK concentration measured. provided.